CLINICAL TRIAL: NCT04347993
Title: Real World Observational Database for COVID-19 Treatment and Outcomes
Brief Title: A Prospective "Universal" Observational Database for COVID-19
Status: Completed | Type: Observational
Sponsor: Hackensack Meridian Health (Other)
Responsible Party: Sponsor
Other Study IDs: Pro2020-0342
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Results first posted 2024-09-03 (Actual); Last update posted 2024-09-03 (Actual); Status verified 2024-04

CONDITIONS: COVID-19
Keywords: Coronavirus; Covid19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Coronavirus Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Hackensack Meridian Health Universal Observational COVID-19, a descriptive observational database, is a multi-center initiative collecting data throughout the Hackensack Meridian Health Network (HMH). HMH utilizes the EPIC system at most of the facilities, which will serve as the primary data source. The database will be designed within the REDCap system. A de-identified dataset will be sent to COTA for primary statistical analysis as requested by the research teams.

DETAILED DESCRIPTION:
The principle objective of this observational database is to build research-grade real world data that will serve as platform to advance the scientific understanding and clinical care of patients with COVID-19.

1. Demographic, diagnostic, treatment and outcome data from centers throughout the Hackensack Meridian Health Network will be abstracted from the electronic health records of patients with confirmed or suspected COVID-19. This will be purely observational and no direction as to the care of the patient will be performed as part of this effort.

1a. Data points to be collected will include, but are not limited to: age, gender, zip code, prior evaluation for COVID-19, tobacco history, race, site of care, healthcare worker, nursing home care, visits to ER, presenting features of fever/ cough/ dyspnea/ gastrointestinal/ mental status changes, days of symptoms, comorbidities, uses of antihypertensives, duration of hospitalization/ icu care, presenting laboratory functions, presenting vital signs, need for oxygen support, dialysis/ ecmo use, treatment with hydroxychloroquine/ azithromycin/ remdesevir/ tociluzimab/ anti-inflammatory agents, arrhythmias/ QTc prolongation, enrollment on clinical trial, positive cultures, survival and cause of death. Additional data points will be added as needed.

2. The data will be entered into a central "Universal" database hosted within the REDCap system (HIPAA compliant, secure, access only per HMH research approval)

3. A de-identified dataset will be sent to COTA for primary statistical analysis as requested by the research teams. COTA will also make available a data/analytic visualization tool (hosted on Tableau) for analysis by primary investigators.

4. Additional data points and analysis may be added to the Universal database as requested by HMH investigators with IRB approval. De-identified data may also be sent directly to HMH investigators for their own analysis with IRB approval of their projects 5. Data will be made available to governmental agencies as requested.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed or suspected COVID-19
* Data available via the EPIC system
* NO age restriction
* NO pregnancy restrictions

Exclusion Criteria:

* Patients on a clinical trial in which the treatment is blinded may be included in the database, however the study medication or treatment will be noted as "experimental" and not reported individually. NO efforts to "break" randomization or blinding will be permitted
* Patients may refuse to be tracked in the database and/or participate in this observational study. Given the lack of active "study" procedures in this observational database, formal informed consent is not required

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with confirmed or suspected COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 4588 (Actual)
Dates: Start 2020-03-27 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Ip, MD, Principal Investigator — Hackensack Meridian Health
Locations (1):
- Hackensack Meridian Health - John Theurer Cancer Center, Hackensack, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Derived] Berry DA, Ip A, Lewis BE, Berry SM, Berry NS, MrKulic M, Gadalla V, Sat B, Wright K, Serna M, Unawane R, Trpeski K, Koropsak M, Kaur P, Sica Z, McConnell A, Bednarz U, Marafelias M, Goy AH, Pecora AL, Sawczuk IS, Goldberg SL. Development and validation of a prognostic 40-day mortality risk model among hospitalized patients with COVID-19. PLoS One. 2021 Jul 30;16(7):e0255228. doi: 10.1371/journal.pone.0255228. eCollection 2021. PMID 34329317
- [Derived] Biran N, Ip A, Ahn J, Go RC, Wang S, Mathura S, Sinclaire BA, Bednarz U, Marafelias M, Hansen E, Siegel DS, Goy AH, Pecora AL, Sawczuk IS, Koniaris LS, Simwenyi M, Varga DW, Tank LK, Stein AA, Allusson V, Lin GS, Oser WF, Tuma RA, Reichman J, Brusco L Jr, Carpenter KL, Costanzo EJ, Vivona V, Goldberg SL. Tocilizumab among patients with COVID-19 in the intensive care unit: a multicentre observational study. Lancet Rheumatol. 2020 Oct;2(10):e603-e612. doi: 10.1016/S2665-9913(20)30277-0. Epub 2020 Aug 14. PMID 32838323
- [Derived] Ip A, Berry DA, Hansen E, Goy AH, Pecora AL, Sinclaire BA, Bednarz U, Marafelias M, Berry SM, Berry NS, Mathura S, Sawczuk IS, Biran N, Go RC, Sperber S, Piwoz JA, Balani B, Cicogna C, Sebti R, Zuckerman J, Rose KM, Tank L, Jacobs LG, Korcak J, Timmapuri SL, Underwood JP, Sugalski G, Barsky C, Varga DW, Asif A, Landolfi JC, Goldberg SL. Hydroxychloroquine and tocilizumab therapy in COVID-19 patients-An observational study. PLoS One. 2020 Aug 13;15(8):e0237693. doi: 10.1371/journal.pone.0237693. eCollection 2020. PMID 32790733

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Confirmed or Suspected COVID-19: Confirmed or suspected COVID-19 with data available via the EPIC system. There are no age restrictions or pregnancy restrictions
Period: Overall Study
Arm/Group | Patients With Confirmed or Suspected COVID-19
Started | 4588
Completed | 4588
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With Confirmed or Suspected COVID-19: Confirmed or suspected COVID-19 Data available via the EPIC system
Arm/Group | Patients With Confirmed or Suspected COVID-19
Number analyzed (Participants) | 4588
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Due to the nature of the retrospective study, not all baseline measures were available in the electronic medical record for all participants.
  years
    number analyzed (Participants) | 4522
    (all) | 60.43 (18.13)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to the nature of the retrospective study, not all baseline measures were available in the electronic medical record for all participants.
  Participants
    number analyzed (Participants) | 4523
    Female | 1914
    Male | 2609
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1041
  Not Hispanic or Latino | 2136
  Unknown or Not Reported | 1411
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 175
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 436
  White | 2249
  More than one race | 0
  Unknown or Not Reported | 1728

OUTCOME MEASURES:

1. Primary Outcome: Need for Hospitalization
Description: Number of Participants needing hospitalization
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Confirmed or Suspected COVID-19
Number analyzed (Participants) | 4588
Participants | 3389

2. Primary Outcome: Duration of Hospitalization
Description: The duration of hospitalization is defined as the time in days from the first day of hospitalized to the date of discharge or death. Patients who are not discharged, are alive and still in the hospital on the date of closing follow-up, or lost follow-up on the date of closing follow-up will be considered censored on that date.
Time Frame: 1 Year
Population: Hospitalized Patients
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Patients With Confirmed or Suspected COVID-19
Number analyzed (Participants) | 3010
Days | 8.93 (10.89)

3. Primary Outcome: Need for ICU/Ventilator Support
Description: Rate of ICU/Ventilator Support
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Confirmed or Suspected COVID-19
Number analyzed (Participants) | 4588
Participants | 853

4. Primary Outcome: Duration of Ventilator Support
Description: The duration of Ventilator Support is defined as the time in days from the first day of using mechanical ventilation to the last day of using mechanical ventilation. All evaluable patients will be included and no censoring for this analysis.
Time Frame: 1 Year
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Patients With Confirmed or Suspected COVID-19
Number analyzed (Participants) | 681
Days | 11.39 (10.24)

5. Primary Outcome: Overall Survival Rate
Description: Overall survival will be defined as rate of patients alive at end of follow up
Time Frame: 1 Year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Confirmed or Suspected COVID-19
Number analyzed (Participants) | 4396
Participants | 3463

ADVERSE EVENTS:
Time Frame: Adverse events were collected for 1 year but this is an observational study and there was no intervention introduced for research purposes.
Groups:
- Patients With Confirmed or Suspected COVID-19: Confirmed or suspected COVID-19 included in the COVID-19 Database Data available via the EPIC system
Arm/Group | Patients With Confirmed or Suspected COVID-19
All-Cause Mortality (participants affected / at risk) | 933/4588
Serious Adverse Events (participants affected / at risk) | 933/4588
Other Adverse Events (participants affected / at risk) | 0/4588
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients With Confirmed or Suspected COVID-19 (N=4588)
Death (Investigations) | 933 (933)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/93/NCT04347993/Prot_SAP_000.pdf